CLINICAL TRIAL: NCT06348810
Title: The Effects of Dual-Task Training on Global Cognitive Function, Executive Function, Working Memory, Sleep, Behavioral Disturbances, Balance, and Flexibility for People With Mild Cognitive Impairment and Mild Dementia
Brief Title: Dual-Task Training for People With Mild Cognitive Impairment and Mild Dementia
Acronym: DTT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei Medical University (Other)
Responsible Party: Principal Investigator, Nur Aini, MSc, Taipei Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: DTT2024
Record Dates: First submitted 2024-03-22; First posted 2024-04-05 (Actual); Last update posted 2024-05-29 (Actual); Status verified 2024-05

CONDITIONS: Dementia; Mild Cognitive Impairment; Older Adult
Keywords: dual-task training; Dementia; Mild Cognitive Impairment; Older adult; Sleep quality; behavioral disturbance; cognition; balance; flexibility
MeSH Terms: conditions — Dementia; Cognitive Dysfunction; Sleep Initiation and Maintenance Disorders; Mental Disorders | interventions — Cognitive Training

STUDY DESIGN:
Intervention Model Description: eksperimental group receive dual-task training, while control group receive usual care and both conduct at the same time
Who Masked: Outcomes Assessor
Masking Description: Outcomes Assessor will be blind, so they didnt know which is intervention group or control group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Dual-task training (Experimental): Participants in the experimental group will receive dual-task training, which consists of cognitive and motor task carried out at the same time. The length of therapy is 12 weeks; sessions are 3 times per week, each session lasts 45 minutes, and total sessions are 36.
  Interventions: Behavioral: Dual-task training
- Cognitive training (Experimental): Participants in this group receive cognitive training only. The length of therapy is 12 weeks; sessions are 3 times per week, each session lasts 45 minutes, and total sessions are 36.
  Interventions: Behavioral: Cognitive training
- Motor training (Experimental): Participants in this group receive motor training only. The length of therapy is 12 weeks; sessions are 3 times per week, each session lasts 45 minutes, and total sessions are 36.
  Interventions: Behavioral: Motor training
- Usual (Active Comparator): Participants in this group receive usual care provided by the nursing home staff, which typically includes assistance with activities of daily living, medication management, and social activities. They do not receive the structured physical exercise program.
  Interventions: Other: Usual care

INTERVENTIONS:
Behavioral: Dual-task training — The dual-task training is a combination of cognitive tasks and motor tasks which is done simultaneously or at the same time.
  Other Names: combination of motor and cognitive task
  Arms: Dual-task training
Behavioral: Cognitive training — Participants only receive cognitive tasks
  Arms: Cognitive training
Behavioral: Motor training — Participants only receive motor tasks
  Arms: Motor training
Other: Usual care — assist participants with activities of daily living, medication management, and social activities (such as singing, watching television).
  Other Names: Routine care
  Arms: Usual

SUMMARY:
Evidence shows that people with dementia have a higher prevalence of sleep disturbance, cognitive decline, behavioral disturbance, and experience motor dysfunction. These symptoms are interrelated. However, few randomized controlled trial (RCT) studies implement dual-task training for mild cognitive impairment and mild dementia, especially for those who experience sleep problems and behavioral disturbances.

Therefore, this study aims to analyze the effect of dual-task training in improving global cognitive function, executive function, working memory, sleep, behavioral disturbances, balance, and flexibility among people with mild cognitive impairment and mild dementia.

The main questions it aims to answer are:

1. . Does dual-task training affect primary outcomes (global cognitive function, executive function, and working memory)
2. . Does dual-task training affect secondary outcomes (including sleep quality, behavioral disturbances, balance, and flexibility) for people with mild cognitive impairment and mild dementia?"

The length of dual-task training is 12 weeks; sessions are 3 times per week, each session lasts 45 minutes, and total sessions are 36. There are three groups of intervention (dual-task training, cognitive training, and motor training). While the control group receives the usual care. Researchers will compare the experiment and control groups to see the effect of the dual-task training.

DETAILED DESCRIPTION:
Sample size calculation: Investigators use the G*Power sample size calculator under an F test with an analysis of variance based on some criteria, for instance: effect size 0.2 (small), power 80%, four times measurement, four groups (cognitive training, motor training, dual-task training, and control group) and α error probability of 0.05. The sample size from the calculator yields 48 in total, considering 50% attrition rate, finally 72 participants (18 participants for each group) will be recruited.

Sample recruitment: Investigator will use a CONSORT flow diagram to describe the phases of this study. A purposive sampling technique will be used in this study to specifically select the nursing home. Following this, eligibility interviews and screening test using MMSE (The Mini Mental State Examination) and The Clinical Dementia Rating (CDR) will be used to recruit participants. The participants will be recruited in this study CDR score varies from 1 to 4, and MMSE >=18. Other inclusion criteria are complain of conscious cognitive decline, participate voluntarily and sign informed consent. However, potential participants will be excluded if they diagnosed with moderate or severe dementia, those who have received cognitive training or motor training within six months, people with severe sensory function impairment (such as vision, hearing), and with limited mobility, such as those using wheelchairs or four-legged walking aids.

Randomization and Blinding: The allocation of the group to be either the experimental (dual-task training group, cognitive training group, motor training group) or control group will be conducted using permuted block randomization design with a block size of four. Randomization was carried out using a web-based randomization tool by a third party who was not involved in the intervention team. To ensure the allocation concealment, investigators use SNOSE principle (sequentially numbered, opaque, sealed envelopes), and randomization code will not be released until the participant or interventionist has started the trial. This study adopts a single-blind approach, by blinding data collector.

Baseline Data Collection Procedure: Participants who meet the inclusion criteria and agree to participate, will be requested to complete a sociodemographic characteristic questionnaire and the seven outcome measures. However, the completion of the seven outcome measures will be conducted in two days to avoid boredom among the participants. In the first period, a sociodemographic questionnaire, WCST, DS, NPI-Q will be completed. The PSQI, ISI, SFBBS, Chair sit-and-reach test (CSR) and Back scratch test completion will be conducted later in the second day at a time agreed upon by the researcher and participants.

Intervention delivery: 1). The dual-task training is a combination of cognitive tasks and motor tasks. Motor task consist of six components, including: strength, balance, agility, gait, aerobic capacity, and flexibility. Whereas Cognitive task consists of four cognitive domains: attention, executive function, learning and memory, language, and perception motor. Both component will be delivered simultaneously or at the same time, and will be delivered in a group format, consisting of 8 to 10 participants for each group. The length of therapy is 12 weeks; sessions are 3 times per week, each session lasts 45 minutes (20 minutes first: cognitive tasks and motor tasks, 5 minutes break time (at this time, participants will be given drink and snack), 20 minutes second: cognitive tasks and motor tasks), and total sessions are 36. In this study, only one interventionist (the principal investigator) from the research team will deliver the intervention sessions. The detail description of each session are below: session 1-6: Participants initially receive one of two tasks (either a cognitive or motor task) and undergo training for each individually; session 7-12: participants receive cognitive and motor task at the same time; session 13-18: repetition of sessions 7 to 12, and session 19-36 are repetition from session 1 to 18. 2). Cognitive training= in this group, participants only receive cognitive training. 3). Motor training= in this group, participants only receive motor training. The duration are same with dual-task training.

Outcomes: The primary outcomes of this study are global cognitive function, executive function, and working memory. Global cognitive is measured using MMSE that consists of five domains. MMSE 0-17 scores indicating severe cognitive impairment, 18-23 mild cognitive impairment, and 24-30 as normal (no cognitive impairment). MMSE was valid and had reliability of 0.763. Executive function in this study will measure using the Wisconsin card sort test (WCST), which has satisfactory reliability and validity for measuring executive function, possessing a split-half reliability of 0.89-0.93 for older adults and test-retest reliability of 0.76. Working memory is measured using a Digit span (DS) test that comprises both digit forward (16 points) and digit backward (14 points). The secondary outcomes of this study are sleep quality, behavioral disturbance, balance, and flexibility. Sleep quality is measured using the Pittsburgh Sleep Quality Index (PSQI) and Insomnia Severity Index (ISI). Behavioral disturbance will be assessed with the Neuropsychiatric Inventory-Questionnaire (NPI-Q). Balance is measured with the Short Form Berg Balance Scale (SFBBS), and flexibilty using flexibility using the Chair sit-and-reach test (CSR) and Back scratch test.

Post-test and Follow-up Data Collection Procedure Participants will be requested to complete questionnares consist of: MMSE, WCST, DS, PSQI, ISI, NPI-Q, SFBBS, Chair sit-and-reach test (CSR) and Back scratch test, in the middle session of the intervention (week 6, after session 18), after intervention completed (week 12, 1 month follow-up time (week 16, measured from baseline)

Statistical analysis: The collected data will be analyzed using IBM SPSS for Windows version 23 and assumed a statistical significance level of p ≤ 0.05. Data consistency checks will be conducted to verify the reliability of the data collected. Descriptive statistics (frequency, percentage, mean, and standard deviation) will be used to summarize the characteristics of the participants and the outcomes. To compare the baseline group differences, investigators will use Chi-square or Fisher exact tests for categorical data, and independent t-tests for continuous data with normal distribution. The generalized estimating equation (GEE) test is used for analyze main outcome with follow the intention-to-treat (ITT) analysis principle, and this test can handle missing data, so no need imputation for missing data.

Interim Analysis and Stopping Guideline: During the study and subsequent follow-up data collection, investigators do not expect any issues that would be harmful to the participants. Investigators have no established termination criteria, and investigators do not plan to perform interim analyses before the follow-up data collection is completed.

ELIGIBILITY:
Inclusion Criteria:

* Older adult >= 60 years and able to communicate
* CDR score range from 1 to 4
* MMSE score >= 18
* Complain of conscious cognitive decline.
* Participate voluntarily and sign informed consent.

Exclusion Criteria:

* Diagnosed with moderate or severe dementia.
* Received cognitive training or motor training within six months.
* Severe sensory function impairment (such as vision, and hearing).
* Have limited mobility, such as those using wheelchairs or four-legged walking aids.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 72 (Estimated)
Dates: Start 2024-07-01 (Estimated); Primary Completion 2024-12-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Global cognitive function | baseline, week 6, week 12, week 16
  measured using MMSE that consists of five domains including orientation to time (5 points), orientation to place (5 points), registration (3 points), attention and calculation (5 points), recall (3 points), and language (9 points), ranges from 0 to 30. MMSE 0-17 scores indicating severe cognitive impairment, 18-23 mild cognitive impairment, and 24-30 as normal (no cognitive impairment).
Executive function | baseline, week 6, week 12, week 16
  measured with the Wisconsin card sort test (WCST). The result of the test is then categorized including: 1). number of completed categories (NCC), 2). total number of errors, 3). perseverative response (PR), 4). perseverative errors, 5). non-perseverative errors (NEs), 6). conceptual level responses (CLRs), 7). failure to maintain set, and 8). trials to complete the first category
Working memory | baseline, week 6, week 12, week 16
  measured using a Digit span (DS) test that comprises both digit forward (16 points) and digit backward (14 points). In the DS forward, the participant had to listen to a digit span that kept to the speed of one digit per second and repeat it forward. In contrast, to DS forward, in the DS backward, the participant had to listen and repeat the span backward. Span was taken as the maximum length if performed without error. However, if participants answered wrong 2 times consequently, the task ended and the number of correct answers was calculated as a score

SECONDARY OUTCOMES:
Sleep Quality | baseline, week 6, week 12, week 16
  Sleep Quality is measured using two instruments. First: Pittsburgh Sleep Quality Index (PSQI). This instrument consists of a 19-item self-rated questionnaire to assess sleep quality during the last month, which includes seven domains, i.e., subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleeping medication, and daytime dysfunction. The score for each domain ranges from 0 to 3, and the total PSQI score ranges from 0 to 21. PSQI score of > 5 indicate poor sleep quality.
  Second: Insomnia Severity Index (ISI). The insomnia severity index is a 7-item self-report questionnaire assessing insomnia's nature, severity, and impact in the past two weeks. The total score is interpreted as follows: absence of insomnia (0-7), sub-threshold insomnia (8-14), moderate insomnia (15-21), and severe insomnia (22-28)
Behavioral disturbance | baseline, week 6, week 12, week 16
  Behavioral disturbance, also known as behavioral and psychological symptoms of dementia (BPSD) or neuropsychiatric symptoms. Behavioral disturbances can be grouped into four categories: mood disorders (such as depression, anxiety, apathy, and euphoria); sleep disorders (such as insomnia, hypersomnia, and night-day reversal); psychotic symptoms (such as hallucinations and delusions); and agitation (such as pacing, wandering, sexual disinhibition, and aggression). Behavioral disturbance will be assessed using the Neuropsychiatric Inventory-Questionnaire (NPI-Q). A higher score pointed to higher severity of neuropsychiatric symptoms (NPS).
Balance | baseline, week 6, week 12, week 16
  measured using the Short Form Berg Balance Scale (SFBBS). Total score varies from 0 to 14. Higher scores indicate better balance and lower risk of falling
Flexibility | baseline, week 6, week 12, week 16
  Flexibility is measured through two ways. The first test is the Chair sit-and-reach test (CSR). CSR is used to measure hamstring flexibility. Participants were instructed to reach down the extended leg in an attempt to touch the toes. The middle of the toe at the end of the shoe represented a "zero" score. Reaches short of the toes were recorded as minus scores, and reaches beyond the toes were recorded as plus scores.
  The second test is Back scratch test, used to measure upper body and shoulder flexibility. The participants started the test by standing upright, placing one arm/hand on the lower back, and moving it up the spine toward their head. The gap between the fingertips of the long fingers of both hands was measured to the nearest half cm. The results were recorded in the nearest half cm, as back scratch right arm and left arm over, with positive numbers as long as the fingers overlapped and with negative numbers if the fingers did not meet.

CONTACTS AND LOCATIONS:
Overall Officials: Nur Aini, MSc, Principal Investigator — School of Nursing, College of Nursing, Taipei Medical University
Locations (1):
- Nursing Home, Malang, East Java, Indonesia

IPD SHARING:
Plan to Share IPD: Yes
Particular data will be shared: Individual participant data that underlie the results reported in this article, after identification (text, tables, figures, and appendices).
Supporting Information: Study Protocol
Time Frame: Beginning 6 months and ending 36 months following article publication.
Access Criteria: Investigators whose proposed use of the data has been approved by an independent review committee ("learned intermediary") identified for this purpose.

REFERENCES:
- [Result] Baltaci G, Un N, Tunay V, Besler A, Gerceker S. Comparison of three different sit and reach tests for measurement of hamstring flexibility in female university students. Br J Sports Med. 2003 Feb;37(1):59-61. doi: 10.1136/bjsm.37.1.59. PMID 12547745
- [Result] Abbas-Zadeh M, Hossein-Zadeh GA, Vaziri-Pashkam M. Dual-Task Interference in a Simulated Driving Environment: Serial or Parallel Processing? Front Psychol. 2021 Jan 12;11:579876. doi: 10.3389/fpsyg.2020.579876. eCollection 2020. PMID 33584415
- [Result] Ambrogio F, Martella LA, Odetti P, Monacelli F. Behavioral Disturbances in Dementia and Beyond: Time for a New Conceptual Frame? Int J Mol Sci. 2019 Jul 25;20(15):3647. doi: 10.3390/ijms20153647. PMID 31349706
- [Result] Bayot M, Dujardin K, Tard C, Defebvre L, Bonnet CT, Allart E, Delval A. The interaction between cognition and motor control: A theoretical framework for dual-task interference effects on posture, gait initiation, gait and turning. Neurophysiol Clin. 2018 Dec;48(6):361-375. doi: 10.1016/j.neucli.2018.10.003. Epub 2018 Oct 26. PMID 30487064
- [Result] Buysse DJ, Reynolds CF 3rd, Monk TH, Berman SR, Kupfer DJ. The Pittsburgh Sleep Quality Index: a new instrument for psychiatric practice and research. Psychiatry Res. 1989 May;28(2):193-213. doi: 10.1016/0165-1781(89)90047-4. PMID 2748771
- [Result] Chiu HL, Chan PT, Kao CC, Chu H, Chang PC, Hsiao SS, Liu D, Chang WC, Chou KR. Effectiveness of executive function training on mental set shifting, working memory and inhibition in healthy older adults: A double-blind randomized controlled trials. J Adv Nurs. 2018 May;74(5):1099-1113. doi: 10.1111/jan.13519. Epub 2018 Jan 24. PMID 29288507
- [Result] Kuan YC, Huang LK, Wang YH, Hu CJ, Tseng IJ, Chen HC, Lin LF. Balance and gait performance in older adults with early-stage cognitive impairment. Eur J Phys Rehabil Med. 2021 Aug;57(4):560-567. doi: 10.23736/S1973-9087.20.06550-8. Epub 2020 Dec 1. PMID 33258361
- [Result] Tzeng RC, Yang YW, Hsu KC, Chang HT, Chiu PY. Sum of boxes of the clinical dementia rating scale highly predicts conversion or reversion in predementia stages. Front Aging Neurosci. 2022 Sep 23;14:1021792. doi: 10.3389/fnagi.2022.1021792. eCollection 2022. PMID 36212036
- [Result] Yang HL, Chu H, Kao CC, Chiu HL, Tseng IJ, Tseng P, Chou KR. Development and effectiveness of virtual interactive working memory training for older people with mild cognitive impairment: a single-blind randomised controlled trial. Age Ageing. 2019 Jul 1;48(4):519-525. doi: 10.1093/ageing/afz029. PMID 30989165
- [Result] Musa G, Henriquez F, Munoz-Neira C, Delgado C, Lillo P, Slachevsky A. Utility of the Neuropsychiatric Inventory Questionnaire (NPI-Q) in the assessment of a sample of patients with Alzheimer's disease in Chile. Dement Neuropsychol. 2017 Apr-Jun;11(2):129-136. doi: 10.1590/1980-57642016dn11-020005. PMID 29213504